CLINICAL TRIAL: NCT01980251
Title: Delirium, Electroencephalographic Alterations and Cortical Spreading Depression in Critical Illness
Brief Title: Delirium, Electroencephalographic Alterations and Cortical Spreading Depression (CSD) in Critical Illness
Status: Completed | Type: Observational
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Rikke Malte Nielsen, M.D., M.D., Glostrup University Hospital, Copenhagen
Other Study IDs: Delirium and cEEG
Record Dates: First submitted 2013-10-24; First posted 2013-11-08 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Delirium
Keywords: Delirium, electroencephalography, CSD
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood, cerebrospinalfluid, urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Delirium in the intensive care unit is an acutely developed brain dysfunction affecting up to 80 % of patients. It is associated with significantly increased morbidity and mortality during admission and post-discharge. The mechanism behind the condition is poorly understood but assumably multifactorial, and the purpose of this study is to investigate the pathophysiology further.

DETAILED DESCRIPTION:
The pathophysiology behind delirium in critical illness is not clarified but assumed to involve inflammation, changes in cerebral perfusion and neurotransmission, sleep deprivation and the use of i.e. sedatives.

Cortical spreading depression is a phenomenon occuring in critically ill patients with acute cerebral trauma and likely associated with significant secondary neuron damage.

The hypothesis is that

1. Delirium in critically ill patients without acute cerebral damage is a clinical manifestation of cortical spreading depression and can be recorded in a noninvasive direct current-electroencephalography
2. Electroencephalographic alterations or potentially specific signatures occur in delirium and thus, delirium can be predicted by recording continuous alternate current electroencephalography on admission in an ICU

ELIGIBILITY:
Inclusion Criteria:

* expected admission in the ICU >24 hours

Exclusion Criteria:

* Cerebral trauma <6 months
* existing delirium
* severe dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with and without acute cerebral trauma
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The occurence of electroencephalographic alterations and potential electroencephalographic signatures prior to and during delirium in the ICU | 7 days

SECONDARY OUTCOMES:
The occurence of cortical spreading depression in noninvasive direct current-EEG in critically ill patients without acute cerebral trauma | Cortical spreading depression in the ICU

OTHER OUTCOMES:
Comparing electroencephalographic and electrocortical recordings in neurointensive care | Delirium - a clinical manifestation of cortical spreading depression?

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Moller, MD, PhD, Study Director — Department of Neuroanaesthesiology 2093, Rigshospitalet, Denmark
Locations (1):
- Glostrup Hospital, University of Copenhagen, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data analysis is in progress

REFERENCES:
- [Derived] Nielsen RM, Urdanibia-Centelles O, Vedel-Larsen E, Thomsen KJ, Moller K, Olsen KS, Lauritsen AO, Eddelien HS, Lauritzen M, Benedek K. Continuous EEG Monitoring in a Consecutive Patient Cohort with Sepsis and Delirium. Neurocrit Care. 2020 Feb;32(1):121-130. doi: 10.1007/s12028-019-00703-w. PMID 30891696